CLINICAL TRIAL: NCT02363179
Title: Music in Urgent and Emergent Settings (MUES) Trial: Phase Two
Brief Title: Music in the Emergency Department (ED): Phase II
Acronym: MUES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of State Division Of Cultural Affairs (Unknown); National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201500083; 15-8503 (Other Grant/Funding Number: FL DEPT OF STATE DIV OF CULTURAL AFFAIRS)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Music Therapy; Patient Satisfaction
Keywords: Emergency Service, Hospital
MeSH Terms: conditions — Patient Satisfaction; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Music Group (No Intervention): 500 non-intervention patients will be consented to serve as the control group
- Music Intervention Group (Experimental): 500 intervention patients will be consented to participate in the live preferential music intervention
  Interventions: Behavioral: Live preferential music

INTERVENTIONS:
Behavioral: Live preferential music — Live preferential music will be performed for patients in the emergency department.
  Arms: Music Intervention Group

SUMMARY:
The investigators will conduct a prospective quasi-experimental design study of patients in the University of Florida Health Emergency Department. Live preferential music will be performed for patients in the emergency department on alternating days over 20 weeks, and subjects exposed to the music intervention will be matched to a cohort that present to the emergency department on days with no music to assess impact on patient and healthcare provider satisfaction, pain medication utilization, length of stay, and cost of care.

DETAILED DESCRIPTION:
Every year, over 130 million patients access emergency care in the US. Emergency Departments are high stress environments and are one of the significant drivers of high costs in healthcare. The prevalence of anxiety experienced by patients in the emergency department (ED) is abundant and substantial. Anxiety negatively affects the patient, the ED healthcare environment, and ED healthcare staff. Additionally, anxiety routinely results in the administration of medication that would be otherwise unnecessary, and contributes to the overall cost of healthcare and the stress of clinicians, particularly nursing staff. The University of Florida (UF) Department of Emergency Medicine, in partnership with the UF Center for Arts in Medicine, has recently completed phase one, and is proposing phase two, of a three-phase study to assess the impact of live preferential music on emergency department operations, including pain medication utilization and cost of care. The investigators propose to expand on the phase one pilot study to conduct a full randomized controlled study utilizing a group of highly talented musicians to provide live preferential music in our ED and level one trauma center setting. The project, the first systematic investigation of its kind, seeks to demonstrate that live preferential music in an emergency and trauma care setting can positively impact quality and cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Language: english
* Cognitive skill/education: grade 2 reading level or above

Exclusion Criteria:

* Language: Non-english speaking
* Age: Less than 18
* Cognitive skill/education: lower than grade 2 reading level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain Medication Utilization | 20 weeks
  Pain Medication Usage

SECONDARY OUTCOMES:
Cost of Care | 20 weeks
  Assessment of the chart associated cost per patient

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Tyndall, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

REFERENCES:
- [Background] Rothrock SG, Johnson NE. Pain management in the pediatric emergency department. Pediatr Emerg Care. 1989 Dec;5(4):298. No abstract available. PMID 2602211
- [Background] Bengtsson SL, Ullen F, Ehrsson HH, Hashimoto T, Kito T, Naito E, Forssberg H, Sadato N. Listening to rhythms activates motor and premotor cortices. Cortex. 2009 Jan;45(1):62-71. doi: 10.1016/j.cortex.2008.07.002. Epub 2008 Oct 30. PMID 19041965
- [Background] Gallagher LM. The role of music therapy in palliative medicine and supportive care. Semin Oncol. 2011 Jun;38(3):403-6. doi: 10.1053/j.seminoncol.2011.03.010. PMID 21600370
- [Background] Good M. A comparison of the effects of jaw relaxation and music on postoperative pain. Nurs Res. 1995 Jan-Feb;44(1):52-7. PMID 7862546
- [Background] Good M, Stanton-Hicks M, Grass JA, Anderson GC, Lai HL, Roykulcharoen V, Adler PA. Relaxation and music to reduce postsurgical pain. J Adv Nurs. 2001 Jan;33(2):208-15. doi: 10.1046/j.1365-2648.2001.01655.x. PMID 11168704